CLINICAL TRIAL: NCT05376319
Title: A Randomized, Double-Blind, Active Comparator-Controlled Study to Evaluate the Effect of Obinutuzumab Versus Rituximab in PR3-Patients With Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis
Brief Title: PR3-AAV Resilient Remission or PRRR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn by sponsor.
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ulrich Specks, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-012197
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis; ANCA Associated Vasculitis
Keywords: Granulomatosis with Polyangiitis; Microscopic Polyangiitis; PR3-ANCA; ANCA-associated Vasculitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — obinutuzumab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous dose of obinutuzumab (Experimental): Subjects who have clinical diagnoses of either granulomatosis with polyangiitis or microscopic polyangiitis will receive two intravenous doses of obinutuzumab
  Interventions: Drug: Obinutuzumab
- Intravenous dose of rituximab (Active Comparator): Subjects who have clinical diagnoses of either granulomatosis with polyangiitis or microscopic polyangiitis will receive two intravenous doses of rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Obinutuzumab — 1000 mg per infusion given approximately two weeks apart, on day 1 and on day 15
  Arms: Intravenous dose of obinutuzumab
Drug: Rituximab — 1000 mg per infusion given approximately two weeks apart, on day 1 and on day 15
  Arms: Intravenous dose of rituximab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of obinutuzumab for the treatment of proteinase 3 Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis (PR3-AAV).

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the definitions of the Second Chapel Hill Consensus Conference for ANCA-associated vasculitis (either granulomatosis with polyangiitis or microscopic polyangiitis).
* Positivity for ANCA, directed against proteinase-3 (PR3)
* Severe newly-diagnosed disease or severe relapsing disease. Severe relapsing disease is defined as at least one major BVAS/WG item or a score ≥ 3 and the investigator deems standard treatment for severe disease is necessary.
* Minimum BVAS/WG of 3
* Relapsing patients must have B cells detectable in the peripheral blood.
* Patients must have completed COVID19 vaccination (including booster if eligible) at least 4 weeks prior to enrollment with a positive spike protein antibody test result. Patients who have recovered from COVID19 prior to screening with a positive spike protein antibody test result but have not been vaccinated are also eligible.
* Female subjects of childbearing potential who are not sterile must agree to use an acceptable method of contraception for 18 months after the last dose of infusion medication. Male subjects who are not sterile whose female partners are of childbearing potential must agree to use an acceptable method of contraception for 180 days after the last dose of infusion medication.

  * Females of childbearing potential include any female who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (to be considered postmenopausal, the patient must have had amenorrhea for >12 consecutive months).
  * Acceptable methods of contraception include the use of at least two of the following: 1) intrauterine device; 2) hormonal contraceptives for at least 30 days prior to first dose infusion (oral, injectable, implant or ring); 3) barrier contraceptives (condom or diaphragm) with spermicide; or 4) abstinence.

Exclusion Criteria:

* Diagnosis with eosinophilic granulomatosis with polyangiitis (formerly Churg-Strauss syndrome) as defined by the Chapel Hill Consensus Conference.
* Positive serum assays for ANCA directed against myeloperoxidase (MPO-ANCA)
* Non-severe AAV, defined as disease that does not justify treatment with both B cell depletion and a four-month glucocorticoid taper.
* Any of the co-morbidities:

  * Allergies: a history of severe allergic reactions to human or chimeric monoclonal antibodies or murine protein.
  * Infection (systemic): an active systemic infection at screening visit
  * Infection (deep space): have been diagnosed as having a deep-space infection, such as osteomyelitis, septic arthritis, or pneumonia complicated by empyema or lung abscesses, within 6 months prior to the screening visit
  * Infection (blood borne): active hepatitis B or active hepatitis C or a documented history of HIV, hepatitis B, or hepatitis C
  * Infection (history): History of recurrent significant infection or history of recurrent bacterial infections
  * Liver disease: acute or chronic liver disease that is deemed sufficiently severe to impair their ability to participate in the trial.
  * Renal disease: a history of documented anti-glomerular basement membrane disease (anti-GBM disease).
  * Malignancy: Active or history of malignancy in the last 5 years. Individuals with squamous cell or basal cell skin carcinomas and individuals with cervical carcinoma in situ may be enrolled if they have received curative surgical treatment.
  * Active COVID-19 infection.
  * Uncontrolled disease: evidence of glucocorticoid dependent disease (such as asthma, COPD, psoriasis or IBD, etc.) requiring consistently greater than 10 mg of prednisone for disease control which might affect endpoint assessment or,
  * Other uncontrolled diseases, including any uncontrolled psychiatric disorders, drug and alcohol abuse, that could interfere with participation in the trial according to the protocol.
* Diagnosis of human anti-chimeric antibodies (HACA) formation.
* Subjects who are premenopausal and are:

  * Pregnant on the basis of a serum pregnancy test,
  * Breastfeeding, or
  * Do not agree to use effective method(s) of contraception
* Use of prohibited medications: They have used any of the prohibited medication listed in Section 5.9.1.
* Plasma exchange: They have been treated with plasma exchange within the 3 months preceding the screening visit.
* History of intolerance to rituximab or other chimeric monoclonal antibodies (e.g., infliximab).
* Recent vaccination: They have had a live vaccine fewer than 4 weeks (28 days) before or during randomization (vaccination with live vaccine through the end of study participation is contraindicated).
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Exclusion criteria related to laboratory parameters:

  * Bone marrow suppression as evidenced by a total white count < 4 x10 /l, hemoglobin < 7 gm/dl or platelet count < 100,000/μl
  * Aspartate aminotransferase or alanine aminotransferase or amylase > 2.5 times the upper limit of normal, unless attributed to vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Specks, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Dose of Obinutuzumab: Subjects who have clinical diagnoses of either granulomatosis with polyangiitis or microscopic polyangiitis received two intravenous doses of obinutuzumab
  Obinutuzumab: 1000 mg per infusion given approximately two weeks apart, on day 1 and on day 15
- Intravenous Dose of Rituximab: Subjects who have clinical diagnoses of either granulomatosis with polyangiitis or microscopic polyangiitis received two intravenous doses of rituximab
  Rituximab: 1000 mg per infusion given approximately two weeks apart, on day 1 and on day 15
Period: Overall Study
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
Started | 2 | 4
Completed | 0 | 0
Not Completed | 2 | 4
Not completed — Funding termination | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 54 [50 to 58] | 53 [19 to 64] | 53.3 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients to Achieve Both Complete Remission and Seronegativity for ANCA.
Description: Complete remission is defined as a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of 0 without glucocorticoids beyond the prescribed prednisone taper. Seronegativity for ANCA is defined as a negative test for antibodies directed against serine proteinase 3 (i.e., a negative PR3-ANCA assay).
Time Frame: 6 months
Population: Terminated study due lack of funding. Data was not collected nor analyzed due to lack of funding. Only one subject in each arm reached 6 months. Data was not collected nor analyzed for 1 subject in the Intravenous dose of obinutuzumab and 3 subjects in the Intravenous dose of rituximab.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Patients to Achieve Sustained Complete Remission 6 Months
Description: Complete remission is defined as a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of 0 without glucocorticoids beyond the prescribed prednisone taper.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

3. Secondary Outcome: Number of Patients to Achieve Sustained Complete Remission 12 Months
Description: as for outcome 2
Time Frame: 12 months
Population: Terminated study due lack of funding. Data was not collected nor analyzed due to lack of funding. Data was not collected nor analyzed for 2 subjects in the Intravenous dose of obinutuzumab and 4 subjects in the Intravenous dose of rituximab.
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients to Achieve Sustained Complete Remission 18 Months
Description: as for outcome 2
Time Frame: 18 months
Population: as for outcome 3
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study for a total of approximately eighteen months
Arm/Group | Intravenous Dose of Obinutuzumab | Intravenous Dose of Rituximab
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Dose of Obinutuzumab (N=2) | Intravenous Dose of Rituximab (N=4)
Sepsis (Infections and infestations) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Dose of Obinutuzumab (N=2) | Intravenous Dose of Rituximab (N=4)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vaginal Yeast Infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hot Flashes (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Voice loss (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening tinnitus (left ear) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right-sided pleuritic abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bilateral thigh discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral knee ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral ankle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension, grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bilateral peripheral ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was discontinued early due to funding termination by industry sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT05376319/Prot_SAP_000.pdf